CLINICAL TRIAL: NCT06151704
Title: The Effect of High-power Laser Therapy on Pain, Functional Disability, Range of Motion and Pressure Pain Threshold in Subjects With Radicular Low Back Pain Due to Intervertebral Disc Herniation: A Double-blind Randomised Controlled Trial
Brief Title: The Effect of High-power Laser Therapy on Pain, Functional Disability, Range of Motion and Pressure Pain Threshold in Subjects With Radicular Low Back Pain Due to Intervertebral Disc Herniation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IR.IUMS.REC.1401.089; IRCT20220410054486N1 (Registry Identifier: Iranian Rigestry of Clinical Trials)
Record Dates: First submitted 2023-11-20; First posted 2023-11-30 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2023-11

CONDITIONS: Radiculopathy, Lumbosacral Region; Radiculopathy Lumbar
Keywords: Low back pain; Disc herniation; Sciatica; High intensity laser therapy; Pain; Functional disability; Range of motion; Pressure pain threshold
MeSH Terms: conditions — Radiculopathy; Low Back Pain; Intervertebral Disc Displacement; Sciatica; Pain

STUDY DESIGN:
Intervention Model Description: The present study is designed as a randomized, double-blind, controlled clinical trial, with control established through sham treatment. The variable block method, comprising four-letter blocks, will be employed for random allocation. The allocation sequence will be determined using the website Generatorslist.com
Who Masked: Participant, Outcomes Assessor
Masking Description: both the patients and the outcome assessor are blinded to the treatment groups. Initially, the assessor measures the outcomes before the patients are included in the study. The therapist then administers the treatments for both groups, with the assessor remaining unaware of the specific treatment throughout the study. Patients are first provided with a comprehensive explanation that the study is a clinical trial consisting of two groups, and they will be randomly assigned to either the intervention group or the control group. All patients are required to wear a protective blindfold during treatment due to the laser procedure. To create authentic therapeutic conditions for the placebo group, the patient is positioned prone with a pillow under their abdomen and wears a protective blindfold. The only difference is that the laser is turned off, and an audio player simulates the sound of the laser device. Upon completion of the study, the examiner conducts the final evaluation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- True high intensity laser therapy on lumbar region, sciatic, tibial, and peroneal nerves (Experimental): The laser scanner, 50 cm from the skin, will target the area from the 12th ribs to the upper iliac crest, 4.2 cm lateral to the spine. The sciatic, tibial, and peroneal nerves will also be irradiated.
  Interventions: Radiation: High intensity laser therapy; Other: Motor control exercise
- Deactivated high intensity laser therapy, an audio device will mimic the laser's operational sound (Sham Comparator): the laser will remain deactivated, and an audio device will generate a simulation of the operational sound of the device. The subject will also participate in the same foundational treatment regimen involving motor control exercises as the intervention group.
  Interventions: Other: Motor control exercise

INTERVENTIONS:
Radiation: High intensity laser therapy — The subject will receive high-intensity laser therapy in a prone position with a cushion under the abdomen and eye protection. The laser scanner, 50 cm from the skin, will target the area from the 12th ribs to the upper iliac crest, 4.2 cm lateral to the spine. The sciatic, tibial, and peroneal nerves will also be irradiated. A GaAlAs laser device will be used, with a power of 1.6 watts and a wavelength of 808nm. The initial dose will be 10 joules/cm², with an increment of 2 joules after every three sessions. The final dose will be 16 joules/cm².
  Other Names: High power laser
  Arms: True high intensity laser therapy on lumbar region, sciatic, tibial, and peroneal nerves
Other: Motor control exercise — Motor control exercise is defined as an exercise to increase control and coordination of the spine and pelvis. Normally, Motor control exercise increases the weak deep trunk muscles, such as transversus abdominis and multifidus, and reduces the overactive large external trunk muscles, such as rectus abdominal and erector spinae muscles. . All subjects participate in a foundational treatment regimen involving motor control exercises: isolated and combined contractions of the transverse abdominis and multifidus muscles in various positions. Contractions will initially be performed up to a maximum of 10 repetitions per movement, with each contraction sustained for a duration of 10 seconds. Commencing from the third week, the subject should be capable of comfortably executing 10 repetitions, sustaining the contraction for 10 seconds, and progressively increasing the intensity.
  Other Names: Stability exercise

SUMMARY:
Low back pain is the predominant cause of disability on a global scale. In the year 2015, the worldwide point prevalence of activity-limiting low back pain stood at 7·3%, suggesting that at any given moment, 540 million individuals were afflicted. In that same year, low back pain emerged as the primary cause of involuntary labor leave and premature retirement within Europe. In the United States, 44% of patients have utilized their health insurance for low back pain at least once, and 1 to 2% (approximately 3 million individuals) exhibit symptoms of sciatica as a result of a lumbar intervertebral disc herniation.

Given the prevalence of disorders attributable to L4-L5 and L5-S1 intervertebral disc herniation, it is imperative to consider the potential risks associated with both surgical and non-surgical medical interventions, such as corticosteroid injections. Laser therapy emerges as a viable modality within the realm of physical therapy, particularly in the mitigation of inflammation. The modulating effects of laser therapy on inflammation have been documented, with no significant side effects reported thus far. Should the efficacy of laser therapy be substantiated, it could be incorporated into the suite of treatments endorsed by authoritative guidelines pertaining to back pain. Patients afflicted with radicular back pain have been the beneficiaries of assistance from physiotherapists possessing specialized knowledge in effective dosimetry. The objectives of this assistance include the amelioration of pain symptoms, the enhancement of functional indicators, the augmentation of the range of motion, and the modulation of the pressure pain threshold, all without the concern of side effects. Furthermore, adherence to the correct treatment protocol is of paramount importance.

The main objective of this study is to evaluate the effect of active high-power laser compared to sham laser on pain, disability, range of motion, and pressure pain threshold in patients with radicular low back pain due to lumbar intervertebral disc herniation.

DETAILED DESCRIPTION:
Risk factors contributing to discopathy disorders encompass repeated asymmetric bending and straightening, which predominantly inflicts damage to the posterolateral portion of the disc. Age constitutes another significant risk factor, with the highest incidence observed between the ages of 30 to 50 due to the watery intervertebral disc. Malignant changes associated with infection, end-plate defect, disease, herniation, genetics, and lifestyle (such as smoking) can lead to a loss of organization of the annulus fibrosus (as seen in myxomatous disease) and a fibrotic nucleus. One of the principal causes of sciatica symptoms is the presence of inflammatory cytokines at the site of the nerve root. These cytokines are released upon damage to the nucleus pulposus, instigating inflammation throughout the surrounding tissues. Given that the majority of disc herniations occur within the canal, inflammation typically affects the nerve roots as well. Mediators such as TNF α, prostaglandin E2, the interleukin group, and phospholipase A2 are implicated in this process." In a study conducted in 1993 by Olmarker et al., an experiment was performed where a fragment of the nucleus was positioned adjacent to a pig's cauda equina nerve, devoid of any mechanical pressure. The conclusion drawn from this experiment was that radicular pain did not originate from a mechanical phenomenon, but rather it led to a reduction in sensation and a decrease in the nerve rate. In a separate group of pigs, a singular mechanical stress was introduced, and the lack of symptoms was subsequently demonstrated. The observations of both localized and extensive hyperalgesia indicate the possibility of pain sensitization. Certain chronic conditions, such as nonspecific shoulder pain, lower back pain, and upper limb disorders, have shown a heightened sensitivity to nerve touch. It has been proposed that this sensitivity of the nerves can be attributed to peripheral sensitization mechanisms, wherein neurogenic inflammation results in the sensitization of neural mechanoreceptors, also known as nervi-nervorum. Furthermore, central sensitization mechanisms may also play a role in nerve sensitization, where non-noxious stimuli from the mechanoreceptors undergo abnormal processing in the central nervous system.

"Numerous studies have meticulously examined the available treatments for intervertebral disc lesions, encompassing both invasive and non-invasive approaches. Surgical interventions, a common modality, have been thoroughly evaluated. However, it is essential to note that patients who underwent surgery did not experience significantly greater pain relief or a more expedited return to work after a 4-year period compared to those who did not undergo surgery. Another invasive treatment involves the administration of injectable corticosteroids. A systematic review conducted by Yang et al. in 2020 meticulously compared physiotherapy interventions (excluding laser therapy) with epidural corticosteroid injections. Surprisingly, the long-term effects of epidural corticosteroid injections were found to be no more efficacious than those of physiotherapy treatments. In a 2015 study by Johnson et al., the pivotal role of TNF-α and IL-1β was elucidated. While these mediators are indispensable for normal physiological function, excessive secretion can indeed be detrimental. The study underscored the importance of precisely controlling the timing of inflammatory secretions and preventing an unwarranted surge in mediator levels to enhance the effectiveness of future treatments." In a 2015 guideline study of medical interventions, including medication, researchers found insufficient evidence to either accept or reject the effects of NSAIDs, muscle relaxants, oral corticosteroids, analgesics, and neuromodulators. Similarly, in a 2017 study by Ghaseem et al., although the evidence for laser therapy was limited, the guideline recommended the use of lasers for patients with low back pain. A study conducted by Maher et al. in 2004 examined the effectiveness of various physiotherapy treatments in systematic studies. Among these treatments, exercise therapy, laser therapy, and manual therapy were the most effective. However, treatments such as hydrotherapy, traction, magnet, and TENS lacked sufficient evidence. Recent studies by Alayat et al. in 2014 did not accept laser therapy as a standalone treatment; its effectiveness has been described only in combination with other physiotherapy treatments.

"Laser, an acronym for Light Amplification by Stimulated Emission of Radiation, possesses three distinct characteristics in the realm of light: 1) Monochromaticity, 2) Coherence (identical phase), and 3) Collimation (high convergence). In this methodology, light energy is projected onto the tissues of the body and absorbed, thereby stimulating or inhibiting enzymatic activity at the cellular level. This instigates physiological reactions, as well as anti-inflammatory and analgesic processes.

Laser therapy promotes interactions between the nucleus and the cytoplasm by augmenting physiological activity within the cell. Near-infrared wavelengths enhance the production of Adenosine Triphosphate (ATP) and alleviate pain and edema by stimulating Cytochrome c oxidase (CcO) at the mitochondrial level. Post-laser irradiation in tissues, there is an observed increase in the levels of beta-endorphins and morphine-mimetic substances, which are natural analgesics produced by the body.

Furthermore, laser irradiation augments lymph flow, decreases prostaglandin synthesis, mitigates the severity of inflammation, and expedites wound healing by enhancing growth factors and phagocytosis, increasing cytokine secretion, promoting angiogenesis, and stimulating fibroblasts and keratinocytes.

Therapeutic lasers, exhibiting a photobiomodulation effect and utilized for pain reduction, are categorized into two types: Low-Level Laser Therapy (power ranging from 5 to 500 mW) and High-Intensity Laser Therapy (power exceeding 500 mW). Laser power is defined as energy per unit time, hence, the use of a high-power laser enables energy to reach the target tissue in a shorter span of time, rendering it more suitable for the treatment of larger areas.

According to the Arendt-Schulz law, a physiological response is elicited in the target tissue once sufficient energy has been delivered to it. In this context, the parameters of the laser and its therapeutic capabilities are of paramount importance." The objective of this study was to ascertain the impact of high-intensity lasers on patients suffering from lower back pain, accompanied by radicular pain in a lower limb, a condition attributed to intervertebral disc herniation. Existing evidence implies that the chronic stage of intervertebral disc herniation may involve inflammatory factors, which could be a primary cause of lower back pain with radicular pain. Given its anti-inflammatory properties and absence of side effects for the patient, the high-power laser could serve as an effective treatment modality in the realm of physiotherapy for patients experiencing radicular lower back pain. This, however, is contingent on the physiotherapist's understanding of dosimetry and the aim of specific dosing therapy. Conversely, the dearth of current research on high-intensity lasers and their impact on lower back pain resulting from intervertebral disc herniation, coupled with diffuse pain in the lower extremities, and the absence of an appropriate treatment protocol, such as the application of high-intensity lasers on pain propagation and proper dosimetry with clinical symptoms, led us to identify a need for community therapy in this study.

The rationale behind selecting exercise therapy as a standard treatment for both groups was the advantageous effects of laser therapy when used in conjunction with exercise therapy. Current studies on the influence of motor control exercises on disc health and on patients with disc herniation suggest that this type of intervention surpasses other exercises (such as strengthening/resistance exercises, cardiovascular, etc.) and other conventional interventions (such as TENS). The treatment plan for patients with disc herniation can have a positive impact on the process of enhancing the reabsorption of herniated disc contents, disc height, disc diffusion rate, and the improvement of radicular symptoms.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of radicular low back pain, originating from an intervertebral disc herniation between the fourth lumbar and first sacral vertebrae, is confirmed by a neurosurgeon
* A minimum of 12 weeks have elapsed since the onset of symptoms. The patient experiences persistent pain or paraesthesia (numbness and/or tingling) in the lower back or both limbs, attributable to the herniation of the lumbar intervertebral disc impinging on the nerve root dermatome
* Magnetic Resonance Imaging (MRI) scans of the patients reveal either protrusion or extrusion disc herniation.

Exclusion Criteria:

* Local or systemic infection, rheumatic disease, diabetes
* Vertebral and sacroiliac joint dysfunction (Gillette test positive)
* Pregnancy
* History of previous surgery in the area
* Patients with MRI of spinal canal stenosis or spondylolisthesis
* Patients with vascular disorders, cancer and tumors and synovial cysts
* History of physiotherapy for at least the last 12 weeks
* sciatic nerve Contusion
* psychiatric illnesses
* Active trigger point of gluteus minimus muscle (diffuse sciatica-like pain)

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2024-12-25 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | This scale will be measured by the assessor prior to the intervention, four weeks after start of treatment, and one month post-treatment. The average pain experienced over the preceding seven days will be recorded as the VAS score
  The Visual Analog Scale, rated from zero (indicating no pain) to 10 (representing the most severe pain conceivable), will be utilized to assess lumbar and affected extremity pain

SECONDARY OUTCOMES:
Functional Disability | This assessment will be conducted by the assessor before the start of treatment, four weeks after start of tratment , and one month post-treatment.
  The functional disability will be evaluated using the validated and reliable Oswestry questionnaire, validated by Mousavi et al. in 2006.
Pressure Pain Threshold | These assessments will be conducted before the start of treatment, four weeks after treatment, and one month post-treatment.
  An algometer will be employed to measure the pressure pain threshold. The algometer will record each point thrice, and the average value per point will be documented. The measurements will be taken at specific points on the body, including 2 and 5 cm lateral to the first and third lumbar vertebrae, 2 cm lateral to the fifth lumbar vertebra, on the common peroneal nerve, tibial nerve, and the sciatic nerve.
Range of Motion | These assessments will be conducted before the start of treatment, four weeks after treatment, and one month post-treatment.
  The active range of motion of the lumbar region (measured using the modified-modified Schubert test) and the Straight Leg Raise (SLR) range of motion of the affected lower limb (measured using a goniometer) will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Seyed Mostafa Teymouri, Msc student, Principal Investigator — Iran University of Medical Sciences; Mohammadreza Pourahmadi, Assistant professor, Study Director — Iran University of Medical Sciences
Locations (1):
- School of Rehabilitation Sciences, Iran University of Medical Sciences, Tehran, Tehran Province, Iran

IPD SHARING:
Plan to Share IPD: Yes
The data sets of this study will be available on a reasonable request to the corresponding author
Time Frame: Starting 6 months after the publication.
Access Criteria: The data will be available for physical therapists working in academic institutions and also clinicians working in the field of musculoskeletal disorders and spine centers. The raw data and results of this study can be used in future relevant systematic reviews. Thus, the raw data and results of this study will be available for researchers working in the field of low back pain. Applicants can contact Seyed Mostafa Teymouri by Email. Email Address:teymouri.seyedmostafa@gmail.com Applicants should explain their project and how the data/documents of the study will be used in their project in detail. Then, the data/documents files will be sent by email to applicants on request. This process may take 10-12 working days

REFERENCES:
- [Background] Hartvigsen J, Hancock MJ, Kongsted A, Louw Q, Ferreira ML, Genevay S, Hoy D, Karppinen J, Pransky G, Sieper J, Smeets RJ, Underwood M; Lancet Low Back Pain Series Working Group. What low back pain is and why we need to pay attention. Lancet. 2018 Jun 9;391(10137):2356-2367. doi: 10.1016/S0140-6736(18)30480-X. Epub 2018 Mar 21. PMID 29573870
- [Background] Knezevic NN, Candido KD, Vlaeyen JWS, Van Zundert J, Cohen SP. Low back pain. Lancet. 2021 Jul 3;398(10294):78-92. doi: 10.1016/S0140-6736(21)00733-9. Epub 2021 Jun 8. PMID 34115979
- [Background] Farfan HF, Cossette JW, Robertson GH, Wells RV, Kraus H. The effects of torsion on the lumbar intervertebral joints: the role of torsion in the production of disc degeneration. J Bone Joint Surg Am. 1970 Apr;52(3):468-97. No abstract available. PMID 5425641
- [Background] Lundon K, Bolton K. Structure and function of the lumbar intervertebral disk in health, aging, and pathologic conditions. J Orthop Sports Phys Ther. 2001 Jun;31(6):291-303; discussion 304-6. doi: 10.2519/jospt.2001.31.6.291. PMID 11411624
- [Background] Beattie PF. Current understanding of lumbar intervertebral disc degeneration: a review with emphasis upon etiology, pathophysiology, and lumbar magnetic resonance imaging findings. J Orthop Sports Phys Ther. 2008 Jun;38(6):329-40. doi: 10.2519/jospt.2008.2768. Epub 2008 Mar 12. PMID 18515962
- [Background] Kawakami M, Matsumoto T, Kuribayashi K, Tamaki T. mRNA expression of interleukins, phospholipase A2, and nitric oxide synthase in the nerve root and dorsal root ganglion induced by autologous nucleus pulposus in the rat. J Orthop Res. 1999 Nov;17(6):941-6. doi: 10.1002/jor.1100170620. PMID 10632462
- [Background] Wanderman RL, Lamer TJ, Wald JT. Myofascial Inflammation Due to Intervertebral Disc Herniation. Pain Med. 2020 Jun 1;21(6):1295-1297. doi: 10.1093/pm/pnaa008. No abstract available. PMID 32053200
- [Background] Risbud MV, Shapiro IM. Role of cytokines in intervertebral disc degeneration: pain and disc content. Nat Rev Rheumatol. 2014 Jan;10(1):44-56. doi: 10.1038/nrrheum.2013.160. Epub 2013 Oct 29. PMID 24166242
- [Background] Burke JG, Watson RW, McCormack D, Dowling FE, Walsh MG, Fitzpatrick JM. Intervertebral discs which cause low back pain secrete high levels of proinflammatory mediators. J Bone Joint Surg Br. 2002 Mar;84(2):196-201. doi: 10.1302/0301-620x.84b2.12511. PMID 11924650
- [Background] Olmarker K, Rydevik B, Nordborg C. Autologous nucleus pulposus induces neurophysiologic and histologic changes in porcine cauda equina nerve roots. Spine (Phila Pa 1976). 1993 Sep 1;18(11):1425-32. PMID 8235812
- [Background] Imamura M, Imamura ST, Kaziyama HH, Targino RA, Hsing WT, de Souza LP, Cutait MM, Fregni F, Camanho GL. Impact of nervous system hyperalgesia on pain, disability, and quality of life in patients with knee osteoarthritis: a controlled analysis. Arthritis Rheum. 2008 Oct 15;59(10):1424-31. doi: 10.1002/art.24120. PMID 18821657
- [Background] Moloney N, Hall T, Doody C. An investigation of somatosensory profiles in work related upper limb disorders: a case-control observational study protocol. BMC Musculoskelet Disord. 2010 Jan 30;11:22. doi: 10.1186/1471-2474-11-22. PMID 20113518
- [Background] Walsh J, Hall T. Reliability, validity and diagnostic accuracy of palpation of the sciatic, tibial and common peroneal nerves in the examination of low back related leg pain. Man Ther. 2009 Dec;14(6):623-9. doi: 10.1016/j.math.2008.12.007. Epub 2009 Feb 6. PMID 19201249
- [Background] Jepsen JR, Laursen LH, Hagert CG, Kreiner S, Larsen AI. Diagnostic accuracy of the neurological upper limb examination I: inter-rater reproducibility of selected findings and patterns. BMC Neurol. 2006 Feb 16;6:8. doi: 10.1186/1471-2377-6-8. PMID 16483371
- [Background] Hall TM, Elvey RL. Nerve trunk pain: physical diagnosis and treatment. Man Ther. 1999 May;4(2):63-73. doi: 10.1054/math.1999.0172. PMID 10509060
- [Background] Quintner JL, Bove GM. From neuralgia to peripheral neuropathic pain: evolution of a concept. Reg Anesth Pain Med. 2001 Jul-Aug;26(4):368-72. doi: 10.1053/rapm.2001.23676. No abstract available. PMID 11464359
- [Background] Fingleton CP, Dempsey L, Smart K, Doody CM. Intraexaminer and interexaminer reliability of manual palpation and pressure algometry of the lower limb nerves in asymptomatic subjects. J Manipulative Physiol Ther. 2014 Feb;37(2):97-104. doi: 10.1016/j.jmpt.2013.12.006. Epub 2014 Jan 3. PMID 24387890
- [Background] O'Connell GD, Leach JK, Klineberg EO. Tissue Engineering a Biological Repair Strategy for Lumbar Disc Herniation. Biores Open Access. 2015 Nov 1;4(1):431-45. doi: 10.1089/biores.2015.0034. eCollection 2015. PMID 26634189
- [Background] Yang S, Kim W, Kong HH, Do KH, Choi KH. Epidural steroid injection versus conservative treatment for patients with lumbosacral radicular pain: A meta-analysis of randomized controlled trials. Medicine (Baltimore). 2020 Jul 24;99(30):e21283. doi: 10.1097/MD.0000000000021283. PMID 32791709
- [Background] Johnson ZI, Schoepflin ZR, Choi H, Shapiro IM, Risbud MV. Disc in flames: Roles of TNF-alpha and IL-1beta in intervertebral disc degeneration. Eur Cell Mater. 2015 Sep 21;30:104-16; discussion 116-7. doi: 10.22203/ecm.v030a08. PMID 26388614
- [Background] Kreiner DS, Hwang SW, Easa JE, Resnick DK, Baisden JL, Bess S, Cho CH, DePalma MJ, Dougherty P 2nd, Fernand R, Ghiselli G, Hanna AS, Lamer T, Lisi AJ, Mazanec DJ, Meagher RJ, Nucci RC, Patel RD, Sembrano JN, Sharma AK, Summers JT, Taleghani CK, Tontz WL Jr, Toton JF; North American Spine Society. An evidence-based clinical guideline for the diagnosis and treatment of lumbar disc herniation with radiculopathy. Spine J. 2014 Jan;14(1):180-91. doi: 10.1016/j.spinee.2013.08.003. Epub 2013 Nov 14. PMID 24239490
- [Background] Qaseem A, Wilt TJ, McLean RM, Forciea MA; Clinical Guidelines Committee of the American College of Physicians; Denberg TD, Barry MJ, Boyd C, Chow RD, Fitterman N, Harris RP, Humphrey LL, Vijan S. Noninvasive Treatments for Acute, Subacute, and Chronic Low Back Pain: A Clinical Practice Guideline From the American College of Physicians. Ann Intern Med. 2017 Apr 4;166(7):514-530. doi: 10.7326/M16-2367. Epub 2017 Feb 14. PMID 28192789
- [Background] Maher CG. Effective physical treatment for chronic low back pain. Orthop Clin North Am. 2004 Jan;35(1):57-64. doi: 10.1016/S0030-5898(03)00088-9. PMID 15062718
- [Background] Alayat MS, Atya AM, Ali MM, Shosha TM. Long-term effect of high-intensity laser therapy in the treatment of patients with chronic low back pain: a randomized blinded placebo-controlled trial. Lasers Med Sci. 2014 May;29(3):1065-73. doi: 10.1007/s10103-013-1472-5. Epub 2013 Nov 2. PMID 24178907
- [Background] Alayat MS, Mohamed AA, Helal OF, Khaled OA. Efficacy of high-intensity laser therapy in the treatment of chronic neck pain: a randomized double-blind placebo-control trial. Lasers Med Sci. 2016 May;31(4):687-94. doi: 10.1007/s10103-016-1910-2. Epub 2016 Feb 25. PMID 26914684
- [Background] Santos Jde O, Oliveira SM, Nobre MR, Aranha AC, Alvarenga MB. A randomised clinical trial of the effect of low-level laser therapy for perineal pain and healing after episiotomy: a pilot study. Midwifery. 2012 Oct;28(5):e653-9. doi: 10.1016/j.midw.2011.07.009. Epub 2011 Oct 5. PMID 21982202
- [Background] Ezzati K, Fekrazad R, Raoufi Z. The Effects of Photobiomodulation Therapy on Post-Surgical Pain. J Lasers Med Sci. 2019 Spring;10(2):79-85. doi: 10.15171/jlms.2019.13. Epub 2019 Feb 25. PMID 31360374
- [Background] Kozanoglu E, Basaran S, Paydas S, Sarpel T. Efficacy of pneumatic compression and low-level laser therapy in the treatment of postmastectomy lymphoedema: a randomized controlled trial. Clin Rehabil. 2009 Feb;23(2):117-24. doi: 10.1177/0269215508096173. PMID 19164399
- [Background] Zati A, Valent A. Physical therapy: new technologies in rehabilitation medicine (translated to English). Edizioni Minerva Medica. 2006;2006:162-85.
- [Background] Alayat MSM, Alshehri MA, Shousha TM, Abdelgalil AA, Alhasan H, Khayyat OK, Al-Attar WS. The effectiveness of high intensity laser therapy in the management of spinal disorders: A systematic review and meta-analysis. J Back Musculoskelet Rehabil. 2019;32(6):869-884. doi: 10.3233/BMR-181341. PMID 30932879
- [Background] Ackermann G, Hartmann M, Scherer K, Lang EW, Hohenleutner U, Landthaler M, Baumler W. Correlations between light penetration into skin and the therapeutic outcome following laser therapy of port-wine stains. Lasers Med Sci. 2002;17(2):70-8. doi: 10.1007/s101030200013. PMID 12111589
- [Background] Jacobsen HE, Khan AN, Levine ME, Filippi CG, Chahine NO. Severity of intervertebral disc herniation regulates cytokine and chemokine levels in patients with chronic radicular back pain. Osteoarthritis Cartilage. 2020 Oct;28(10):1341-1350. doi: 10.1016/j.joca.2020.06.009. Epub 2020 Jul 9. PMID 32653386
- [Background] Pedersen LM, Schistad E, Jacobsen LM, Roe C, Gjerstad J. Serum levels of the pro-inflammatory interleukins 6 (IL-6) and -8 (IL-8) in patients with lumbar radicular pain due to disc herniation: A 12-month prospective study. Brain Behav Immun. 2015 May;46:132-6. doi: 10.1016/j.bbi.2015.01.008. Epub 2015 Jan 31. PMID 25653193
- [Background] de Lima FM, Bjordal JM, Albertini R, Santos FV, Aimbire F. Low-level laser therapy (LLLT) attenuates RhoA mRNA expression in the rat bronchi smooth muscle exposed to tumor necrosis factor-alpha. Lasers Med Sci. 2010 Sep;25(5):661-8. doi: 10.1007/s10103-010-0766-0. PMID 20393772
- [Background] de Lima FM, Villaverde AB, Albertini R, Correa JC, Carvalho RL, Munin E, Araujo T, Silva JA, Aimbire F. Dual Effect of low-level laser therapy (LLLT) on the acute lung inflammation induced by intestinal ischemia and reperfusion: Action on anti- and pro-inflammatory cytokines. Lasers Surg Med. 2011 Jul;43(5):410-20. doi: 10.1002/lsm.21053. PMID 21674546
- [Background] Nambi G. Does low level laser therapy has effects on inflammatory biomarkers IL-1beta, IL-6, TNF-alpha, and MMP-13 in osteoarthritis of rat models-a systemic review and meta-analysis. Lasers Med Sci. 2021 Apr;36(3):475-484. doi: 10.1007/s10103-020-03124-w. Epub 2020 Aug 24. PMID 32833088
- [Background] Lopes-Martins RAB, Marcos RL, Leal-Junior ECP, Bjordal JM. Low-Level Laser Therapy and World Association for Laser Therapy Dosage Recommendations in Musculoskeletal Disorders and Injuries. Photomed Laser Surg. 2018 Sep;36(9):457-459. doi: 10.1089/pho.2018.4493. No abstract available. PMID 30188251
- [Background] Searle A, Spink M, Ho A, Chuter V. Exercise interventions for the treatment of chronic low back pain: a systematic review and meta-analysis of randomised controlled trials. Clin Rehabil. 2015 Dec;29(12):1155-67. doi: 10.1177/0269215515570379. Epub 2015 Feb 13. PMID 25681408
- [Background] Franca FJR, Callegari B, Ramos LAV, Burke TN, Magalhaes MO, Comachio J, CarvalhoSilva APMC, Almeida GPL, Marques AP. Motor Control Training Compared With Transcutaneous Electrical Nerve Stimulation in Patients With Disc Herniation With Associated Radiculopathy: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2019 Mar;98(3):207-214. doi: 10.1097/PHM.0000000000001048. PMID 30247159
- [Background] Owen PJ, Miller CT, Rantalainen T, Simson KJ, Connell D, Hahne AJ, Trudel G, Ford JJ, Belavy DL. Exercise for the intervertebral disc: a 6-month randomised controlled trial in chronic low back pain. Eur Spine J. 2020 Aug;29(8):1887-1899. doi: 10.1007/s00586-020-06379-7. Epub 2020 Mar 24. PMID 32211998
- [Background] Kolu E, Buyukavci R, Akturk S, Eren F, Ersoy Y. Comparison of high-intensity laser therapy and combination of transcutaneous nerve stimulation and ultrasound treatment in patients with chronic lumbar radiculopathy: A randomized single-blind study. Pak J Med Sci. 2018 May-Jun;34(3):530-534. doi: 10.12669/pjms.343.14345. PMID 30034410
- [Background] Chen L, Liu D, Zou L, Huang J, Chen J, Zou Y, Lai J, Chen J, Li H, Liu G. Efficacy of high intensity laser therapy in treatment of patients with lumbar disc protrusion: A randomized controlled trial. J Back Musculoskelet Rehabil. 2018 Feb 6;31(1):191-196. doi: 10.3233/BMR-170793. PMID 28854500
- [Background] Boyraz I, Yildiz A, Koc B, Sarman H. Comparison of high-intensity laser therapy and ultrasound treatment in the patients with lumbar discopathy. Biomed Res Int. 2015;2015:304328. doi: 10.1155/2015/304328. Epub 2015 Mar 25. PMID 25883952
- [Background] de Carvalho ME, de Carvalho RM Jr, Marques AP, de Carvalho Lucio LM, de Oliveira AC, Neto OP, Villaverde AB, de Lima CJ. Low intensity laser and LED therapies associated with lateral decubitus position and flexion exercises of the lower limbs in patients with lumbar disk herniation: clinical randomized trial. Lasers Med Sci. 2016 Sep;31(7):1455-63. doi: 10.1007/s10103-016-2009-5. Epub 2016 Jul 5. PMID 27379776
- [Background] Fiore P, Panza F, Cassatella G, Russo A, Frisardi V, Solfrizzi V, Ranieri M, Di Teo L, Santamato A. Short-term effects of high-intensity laser therapy versus ultrasound therapy in the treatment of low back pain: a randomized controlled trial. Eur J Phys Rehabil Med. 2011 Sep;47(3):367-73. Epub 2011 Jun 8. PMID 21654616
- [Background] Abdelbasset WK, Nambi G, Alsubaie SF, Abodonya AM, Saleh AK, Ataalla NN, Ibrahim AA, Tantawy SA, Kamel DM, Verma A, Moawd SA. A Randomized Comparative Study between High-Intensity and Low-Level Laser Therapy in the Treatment of Chronic Nonspecific Low Back Pain. Evid Based Complement Alternat Med. 2020 Oct 28;2020:1350281. doi: 10.1155/2020/1350281. eCollection 2020. PMID 33178306
- [Background] Ay S, Dogan SK, Evcik D. Is low-level laser therapy effective in acute or chronic low back pain? Clin Rheumatol. 2010 Aug;29(8):905-10. doi: 10.1007/s10067-010-1460-0. Epub 2010 Apr 23. PMID 20414695
- [Background] Gonzalez-Lima F, editor Dose-response effects of low-level light therapy on brain and muscle. Proceeding of the 13th Annual International Conference on Dose-Response Texas: The University of Texas at Austin; 2014.
- [Background] Conte P, Santamato A, Fiore P, Lopresto A, Mazzaracchio M. Treatment of chronic low back pain: back school versus Hilterapia. Energy for health. 2009;3(3):10.
- [Background] Choi HW, Lee J, Lee S, Choi J, Lee K, Kim BK, Kim GJ. Effects of high intensity laser therapy on pain and function of patients with chronic back pain. J Phys Ther Sci. 2017 Jun;29(6):1079-1081. doi: 10.1589/jpts.29.1079. Epub 2017 Jun 7. PMID 28626329
- [Background] Zahra ALT, Alhabeel M. Laser Dental Treatment Techniques. 2019. p. 2-16.
- [Background] World Association of Laser Therapy (WALT). Standards for the design and conduct of systematic reviews with low-level laser therapy for musculoskeletal pain and disorders. Photomed Laser Surg. 2006 Dec;24(6):759-60. doi: 10.1089/pho.2006.24.759. No abstract available. PMID 17199478
- [Background] Govind J. Lumbar radicular pain. Aust Fam Physician. 2004 Jun;33(6):409-12. PMID 15253601
- [Background] Alain Y. Belanger therapeutic electrophysical agents: evidence behind practice. Philadelphia, PA: Lippincott Williams & Wilkins; 2015.
- [Background] Krusen FH, Kottke FJ, Ellwood PM. Handbook of physical medicine and rehabilitation: WB Saunders Company; 1971.
- [Background] Williams ACC, Craig KD. Updating the definition of pain. Pain. 2016 Nov;157(11):2420-2423. doi: 10.1097/j.pain.0000000000000613. No abstract available. PMID 27200490
- [Background] Leonardi M, Bickenbach J, Ustun TB, Kostanjsek N, Chatterji S; MHADIE Consortium. The definition of disability: what is in a name? Lancet. 2006 Oct 7;368(9543):1219-21. doi: 10.1016/S0140-6736(06)69498-1. No abstract available. PMID 17027711
- [Background] Mousavi SJ, Parnianpour M, Mehdian H, Montazeri A, Mobini B. The Oswestry Disability Index, the Roland-Morris Disability Questionnaire, and the Quebec Back Pain Disability Scale: translation and validation studies of the Iranian versions. Spine (Phila Pa 1976). 2006 Jun 15;31(14):E454-9. doi: 10.1097/01.brs.0000222141.61424.f7. PMID 16778675
- [Background] Ylinen J. Pressure algometry. Aust J Physiother. 2007;53(3):207. doi: 10.1016/s0004-9514(07)70032-6. No abstract available. PMID 17899675
- [Background] Vucinic N, Eric M, Tomasevic-Todorovic S, Milekic B. Application of algometry in patients with cervical and lumbar radiculopathy. J Back Musculoskelet Rehabil. 2018;31(3):567-575. doi: 10.3233/BMR-170965. PMID 29526842
- [Background] Gajdosik RL, Bohannon RW. Clinical measurement of range of motion. Review of goniometry emphasizing reliability and validity. Phys Ther. 1987 Dec;67(12):1867-72. doi: 10.1093/ptj/67.12.1867. PMID 3685114
- [Background] Tousignant M, Poulin L, Marchand S, Viau A, Place C. The Modified-Modified Schober Test for range of motion assessment of lumbar flexion in patients with low back pain: a study of criterion validity, intra- and inter-rater reliability and minimum metrically detectable change. Disabil Rehabil. 2005 May 20;27(10):553-9. doi: 10.1080/09638280400018411. PMID 16019864
- [Background] Eloqayli H. Clinical Decision-Making in Chronic Spine Pain: Dilemma of Image-Based Diagnosis of Degenerative Spine and Generation Mechanisms for Nociceptive, Radicular, and Referred Pain. Biomed Res Int. 2018 Dec 17;2018:8793843. doi: 10.1155/2018/8793843. eCollection 2018. PMID 30648110
- [Background] Taradaj J, Rajfur K, Shay B, Rajfur J, Ptaszkowski K, Walewicz K, Dymarek R, Sopel M, Rosinczuk J. Photobiomodulation using high- or low-level laser irradiations in patients with lumbar disc degenerative changes: disappointing outcomes and remarks. Clin Interv Aging. 2018 Aug 21;13:1445-1455. doi: 10.2147/CIA.S168094. eCollection 2018. PMID 30174418
- [Background] Yilmaz M, Tarakci D, Tarakci E. Comparison of high-intensity laser therapy and combination of ultrasound treatment and transcutaneous nerve stimulation on cervical pain associated with cervical disc herniation: A randomized trial. Complement Ther Med. 2020 Mar;49:102295. doi: 10.1016/j.ctim.2019.102295. Epub 2020 Jan 3. PMID 32147037
- [Background] Dayanir IO, Birinci T, Kaya Mutlu E, Akcetin MA, Akdemir AO. Comparison of Three Manual Therapy Techniques as Trigger Point Therapy for Chronic Nonspecific Low Back Pain: A Randomized Controlled Pilot Trial. J Altern Complement Med. 2020 Apr;26(4):291-299. doi: 10.1089/acm.2019.0435. Epub 2020 Feb 5. PMID 32023423
- [Background] Ostelo RW, Deyo RA, Stratford P, Waddell G, Croft P, Von Korff M, Bouter LM, de Vet HC. Interpreting change scores for pain and functional status in low back pain: towards international consensus regarding minimal important change. Spine (Phila Pa 1976). 2008 Jan 1;33(1):90-4. doi: 10.1097/BRS.0b013e31815e3a10. PMID 18165753
- [Background] Koumantakis GA, Watson PJ, Oldham JA. Trunk muscle stabilization training plus general exercise versus general exercise only: randomized controlled trial of patients with recurrent low back pain. Phys Ther. 2005 Mar;85(3):209-25. PMID 15733046
- [Background] Roland M, Waddell G, Klaber-Moffett J, Burton A, Main C. The back book: the best way to deal with back pain: TSO; 2002.
- [Background] Fairbank JC, Pynsent PB. The Oswestry Disability Index. Spine (Phila Pa 1976). 2000 Nov 15;25(22):2940-52; discussion 2952. doi: 10.1097/00007632-200011150-00017. PMID 11074683
- [Background] Yalfani A, Raeisi Z, Koumasian Z. Effects of eight-week water versus mat pilates on female patients with chronic nonspecific low back pain: Double-blind randomized clinical trial. J Bodyw Mov Ther. 2020 Oct;24(4):70-75. doi: 10.1016/j.jbmt.2020.06.002. Epub 2020 Jun 27. PMID 33218568
- [Background] Sawilowsky SS. New effect size rules of thumb. Journal of modern applied statistical methods. 2009;8(2):26.